CLINICAL TRIAL: NCT04608760
Title: Prevention of Acute Pancreatitis After Endoscopic Interventions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Vitebsk State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Interventional
Record Dates: First submitted 2020-10-24; First posted 2020-10-29 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Cholangiolitis; Acute Pancreatitis
Keywords: Cholangiolithiasis, endoscopic, acute pancreatitis, cholangiography
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Meksibel (Active Comparator): Intravenous 0.1 30 minutes before the procedure and 0.1 once a day for 3 days after the procedure
  Interventions: Drug: Meksibel
- Indometacin (Active Comparator): Into the rectum 1 hour before the procedure and 1 candle 1 time a day for 3 days after the procedure
  Interventions: Drug: Meksibel
- Meloksicam (Active Comparator): Intravenous 15 mg 30 minutes before the procedure and 15 mg once a day for 3 days after the procedure
  Interventions: Drug: Meksibel
- Oktride (Active Comparator): Intravenous 3 ml 30 minutes before the procedure and 3 ml once a day for 3 days after the procedure
  Interventions: Drug: Meksibel

INTERVENTIONS:
Drug: Meksibel — 2 ml solution

SUMMARY:
The aim of the study is to develop a method for the prevention of acute pancreatitis after minimally invasive interventions of the bile ducts using a drug regimen.

DETAILED DESCRIPTION:
A prospective, randomized, single-center study is planned to identify the most effective drug regimen in order to prevent the development of acute pancreatitis after transpapillary interventions of the bile ducts.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cholangiolithiasis.
2. Patients with benign formations of the bile ducts.
3. Patients with malignant formations of the bile ducts.
4. Patients with extrahepatic bile duct cysts.
5. Patients with biliary hypertension of unknown etiology.
6. Patients with cholangitis.
7. Patients with extrahepatic bile duct strictures.
8. Patients suffering from oncopathology of the head of the pancreas, complicated by obstructive jaundice.
9. Patients with malignant pathology of the pancreas.
10. Patients with benign pancreatic pathology.

Exclusion Criteria:

1. ASA scale> III (severe concomitant cardiovascular pathology)
2. Severe pathology of the respiratory system.
3. Acute period of myocardial infarction.
4. Acute period of cerebral infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in the level of inflammation and pain, assessment of severity according to the Ranson scale and Krasnogorov at 1 week | 1 week
  Summ points 0 - pancreatitis, 1 - mild pancreatitis, 2 - severe pancreatitis

CONTACTS AND LOCATIONS:
Overall Officials: Yury Arlouski, MD, PhD, Study Chair — Vitebsk State Medical University
Locations (1):
- VSMU, Vitebsk, Belarus